CLINICAL TRIAL: NCT00613171
Title: A Multi-centre, Open-label, Proof of Concept (PoC) Study to Evaluate the Efficacy and Tolerability of STI571 for the Treatment of Fibrosis in Patients With Systemic Sclerosis
Brief Title: Efficacy and Tolerability of STI571 (Imatinib Mesylate) for the Treatment of Fibrosis in Participants With Systemic Sclerosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSTI571E2205
Record Dates: First submitted 2008-01-25; First posted 2008-02-12 (Estimated); Results first posted 2021-05-21 (Actual); Last update posted 2021-07-07 (Actual); Status verified 2021-07

CONDITIONS: Systemic Sclerosis, Scleroderma
Keywords: Systemic sclerosis, scleroderma, fibrosis, STI571, imatinib
MeSH Terms: conditions — Scleroderma, Systemic; Scleroderma, Diffuse; Fibrosis | interventions — Imatinib Mesylate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- ST1571 (Experimental): Participants received ST1571 100 mg tablets, orally, once daily. Initiated at an oral dose of 200 mg/day for 4 weeks then titrated up to 400 mg/day for 2 weeks followed by 600 mg/day until Week 24, if well tolerated.
  Interventions: Drug: STI571

INTERVENTIONS:
Drug: STI571 — STI571 tablets taken orally once a day
  Other Names: Gleevec, Glivec

SUMMARY:
This study investigates the efficacy and safety of STI571 for the treatment of fibrosis in participants with systemic sclerosis. Other purposes of the study were to investigate whether STI571 is effective in improving lung functions and other test results called biomarkers. Whether STI571 is well-absorbed in systemic sclerosis participants' gut was also investigated by testing the drug level in the blood (pharmacokinetics).

ELIGIBILITY:
Inclusion Criteria:

* Male and female participants who are equal to or older than 18 years of age and who have early diffuse cutaneous systemic sclerosis (Disease duration < 18 months from the first non-Raynaud's symptom)
* Participants with a modified Rodnans Skin Score (MRSS) of at least 20 in the absence of trunk involvement or a MRSS of at least 16 in patients with trunk involvement
* Female patients of childbearing potential practicing two acceptable forms of contraception

Exclusion Criteria:

* SSc patients with a MRSS greater than 35
* Concurrent connective tissue diseases other than systemic sclerosis
* Significant pre-existing heart, liver, lungs, digestive system, blood and other diseases, cancer
* Conditions that might mimic the potential side effects of STI571 (blood conditions, liver damage, chronic diarrhea, edema)
* Concurrent medical therapies (or during last 6 weeks before first dosing) that may potentially influence outcome of the study
* Allergic to the study medication
* Pregnancy
* Breast feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2008-01-02 (Actual); Primary Completion 2010-01-13 (Actual); Study Completion 2010-01-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: NOVARTIS, Principal Investigator — Novartis investigator site
Locations (7):
- United States (3):
  - Novartis Investigator Site, Chicago, Illinois
  - Novartis Investigator Site, Baltimore, Maryland
  - Novartis Investigator Site, Boston, Massachusetts
- Novartis Investigator Site, Erlangen, Germany
- Novartis Investigator Site, Florence, Italy
- Novartis Investigator Site, Zurich, Switzerland
- Novartis Investigator Site, London, United Kingdom

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 7 centers in 5 countries from 02 January 2008 to 13 January 2010.
Pre-assignment Details: The study enrolled a total of 27 participants. The study consisted of a treatment period of 24 weeks and a follow-up period of 24 weeks with no study drug.
Groups:
- STI571: Participants received ST1571 100 mg tablets, orally, once daily. Initiated at an oral dose of 200 mg/day for 4 weeks then titrated up to 400 mg/day for 2 weeks followed by 600 mg/day until Week 24, if well tolerated.
Period: Overall Study
Arm/Group | STI571
Started | 27
Completed | 13
Not Completed | 14
Not completed — Adverse Event | 7
Not completed — Withdrawal by Subject | 3
Not completed — Reason not Specified | 4

BASELINE CHARACTERISTICS:
Population: Efficacy analysis set included all participants who received at least one dose of the study drug with at least one post-baseline measurement.
Arm/Group | STI571
Number analyzed (Participants) | 27
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.7 (11.99)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21
  Male | 6

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Modified Rodnan Skin Score (MRSS) at Each Time Point of Analysis
Description: The efficacy of oral STI571 in participants with systemic sclerosis is defined by an improvement in MRSS. Skin thickness was assessed clinically in each of 17 body areas and scored using a 0-3 scale, where 0= normal, 1= mild thickness, 2= moderate thickness, and 3= severe thickness (maximum score 51). A higher score indicates greater severity of the disease.
Time Frame: Baseline, Weeks 2, 4, 6, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, and Week 48/End of Study (EOS)
Population: Efficacy analysis set included all participants who received at least one dose of the study drug with at least one post-baseline measurement. Number analyzed are the number of participants with data available for analyses at given time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | STI571
Number analyzed (Participants) | 27
units on a scale
  Baseline | 25.7 (5.83)
  Week 2 | 6.58 (18.416)
  Week 4 | 5.97 (17.382)
  Week 6 | 8.34 (24.645)
  Week 8: number analyzed (Participants) | 24
  Week 8 | 8.48 (27.096)
  Week 12: number analyzed (Participants) | 18
  Week 12 | 3.34 (27.525)
  Week 16: number analyzed (Participants) | 18
  Week 16 | 12.70 (28.399)
  Week 20: number analyzed (Participants) | 18
  Week 20 | 12.41 (28.149)
  Week 24: number analyzed (Participants) | 16
  Week 24 | 9.90 (23.675)
  Week 28: number analyzed (Participants) | 14
  Week 28 | -3.17 (19.891)
  Week 32: number analyzed (Participants) | 14
  Week 32 | -5.67 (18.013)
  Week 36: number analyzed (Participants) | 12
  Week 36 | -12.61 (27.383)
  Week 40: number analyzed (Participants) | 12
  Week 40 | -5.23 (27.506)
  Week 44: number analyzed (Participants) | 13
  Week 44 | -13.57 (26.763)
  Week 48/ EOS: number analyzed (Participants) | 13
  Week 48/ EOS | -20.89 (24.946)

2. Primary Outcome: Number of Participants With Adverse Events (AE's) and Serious Adverse Events (SAE's)
Description: An AE is the appearance or worsening of any undesirable sign, symptom, or medical condition occurring after starting the study drug even if the event is not considered to be related to the study drug. An SAE is defined as an event that is fatal or life-threatening, results in persistent or significant disability/incapacity, constitutes a congenital anomaly/birth defect, requires inpatient hospitalization or prolongation of existing hospitalization, is medically significant, i.e., defined as an event that jeopardizes the patient or may require medical or surgical intervention to prevent one of the outcomes listed above.
Time Frame: Baseline to Week 48/EOS
Population: Safety analysis set included all participants who received at least one dose of the study drug with at least one post-baseline measurement.
Measure: Count of Participants; unit: Participants
Arm/Group | STI571
Number analyzed (Participants) | 27
Participants
  Participants Experiencing AE's | 27
  Participants Experiencing SAE's | 5

3. Secondary Outcome: Number of Participants With Non-response, Partial Response, Complete Response, and Remission Assessed by MRSS Values
Description: The following MRSS categories were calculated for up to Week 48: Non-response: a reduction in MRSS <25%, Partial response: a reduction in MRSS between 25-<50%, Complete response: a reduction in MRSS between 50-<80%, Remission: a reduction in MRSS ≥80%.
Time Frame: Weeks 2, 4, 6, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, and Week 48/End of Study (EOS)
Population: Efficacy analysis set included all participants that received at least one dose of the study drug with at least one post-baseline measurement. Number analyzed are the number of participants with data available for analyses at given time points.
Measure: Count of Participants; unit: Participants
Groups:
- STI571: Participants received STI571 100 mg tablets, once daily. Initiated at an oral dose of 200 mg/day for 4 weeks then titrated up to 400 mg/day for 2 weeks followed by 600 mg/day until Week24, if well tolerated.
Arm/Group | STI571
Number analyzed (Participants) | 27
Participants
  Week 2: Non-response | 27
  Week 2: Partial Response | 0
  Week 2: Complete Response | 0
  Week 2: Remission | 0
  Week 4: Non-response | 25
  Week 4: Partial Response | 2
  Week 4: Complete Response | 0
  Week 4: Remission | 0
  Week 6: Non-response | 24
  Week 6: Partial Response | 2
  Week 6: Complete Response | 1
  Week 6: Remission | 0
  Week 8: number analyzed (Participants) | 24
  Week 8: Non-response | 22
  Week 8: Partial Response | 2
  Week 8: Complete Response | 0
  Week 8: Remission | 0
  Week 12: number analyzed (Participants) | 18
  Week 12: Non-response | 15
  Week 12: Partial Response | 3
  Week 12: Complete Response | 0
  Week 12: Remission | 0
  Week 16: number analyzed (Participants) | 18
  Week 16: Non-response | 16
  Week 16: Partial Response | 2
  Week 16: Complete Response | 0
  Week 16: Remission | 0
  Week 20: number analyzed (Participants) | 18
  Week 20: Non-response | 16
  Week 20: Partial Response | 2
  Week 20: Complete Response | 0
  Week 20: Remission | 0
  Week 24: number analyzed (Participants) | 16
  Week 24: Non-response | 15
  Week 24: Partial Response | 1
  Week 24: Complete Response | 0
  Week 24: Remission | 0
  Week 28: number analyzed (Participants) | 14
  Week 28: Non-response | 13
  Week 28: Partial Response | 1
  Week 28: Complete Response | 0
  Week 28: Remission | 0
  Week 32: number analyzed (Participants) | 14
  Week 32: Non-response | 13
  Week 32: Partial Response | 1
  Week 32: Complete Response | 0
  Week 32: Remission | 0
  Week 36: number analyzed (Participants) | 12
  Week 36: Non-response | 9
  Week 36: Partial Response | 3
  Week 36: Complete Response | 0
  Week 36: Remission | 0
  Week 40: number analyzed (Participants) | 12
  Week 40: Non-response | 9
  Week 40: Partial Response | 3
  Week 40: Complete Response | 0
  Week 40: Remission | 0
  Week 44: number analyzed (Participants) | 13
  Week 44: Non-response | 8
  Week 44: Partial Response | 5
  Week 44: Complete Response | 0
  Week 44: Remission | 0
  Week 48/EOS: number analyzed (Participants) | 13
  Week 48/EOS: Non-response | 5
  Week 48/EOS: Partial Response | 8
  Week 48/EOS: Complete Response | 0
  Week 48/EOS: Remission | 0

ADVERSE EVENTS:
Time Frame: Baseline to Week 48/EOS
Description: Safety analysis set included all participants who received at least one dose of the study drug with at least one post-baseline measurement.
Arm/Group | ST1571
All-Cause Mortality (participants affected / at risk) | 0/27
Serious Adverse Events (participants affected / at risk) | 5/27
Other Adverse Events (participants affected / at risk) | 27/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ST1571 (N=27)
Neutropenia (Blood and lymphatic system disorders) | 1
Gastritis erosive (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Face oedema (General disorders) | 1
Generalised oedema (General disorders) | 1
Oedema peripheral (General disorders) | 1
Neutropenic infection (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 1
Viral infection (Infections and infestations) | 1
Haematocrit decreased (Investigations) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | ST1571 (N=27)
Anaemia (Blood and lymphatic system disorders) | 6
Leukopenia (Blood and lymphatic system disorders) | 1
Lymphopenia (Blood and lymphatic system disorders) | 2
Thrombocytosis (Blood and lymphatic system disorders) | 1
Cardiac disorder (Cardiac disorders) | 1
Auricular swelling (Ear and labyrinth disorders) | 1
Ear pain (Ear and labyrinth disorders) | 1
Tinnitus (Ear and labyrinth disorders) | 1
Vertigo (Ear and labyrinth disorders) | 1
Eye swelling (Eye disorders) | 1
Eyelid oedema (Eye disorders) | 1
Ocular hyperaemia (Eye disorders) | 1
Abdominal discomfort (Gastrointestinal disorders) | 3
Abdominal distension (Gastrointestinal disorders) | 4
Abdominal pain lower (Gastrointestinal disorders) | 1
Abdominal pain upper (Gastrointestinal disorders) | 3
Constipation (Gastrointestinal disorders) | 3
Diarrhoea (Gastrointestinal disorders) | 7
Diverticulum (Gastrointestinal disorders) | 1
Dry mouth (Gastrointestinal disorders) | 1
Dyspepsia (Gastrointestinal disorders) | 4
Faeces discoloured (Gastrointestinal disorders) | 1
Flatulence (Gastrointestinal disorders) | 3
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1
Gingival pain (Gastrointestinal disorders) | 1
Hypoaesthesia oral (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 14
Tongue dry (Gastrointestinal disorders) | 1
Toothache (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 5
Face oedema (General disorders) | 5
Fatigue (General disorders) | 5
Generalised oedema (General disorders) | 1
Influenza like illness (General disorders) | 2
Infusion site ulcer (General disorders) | 1
Oedema (General disorders) | 1
Oedema peripheral (General disorders) | 15
Pyrexia (General disorders) | 1
Herpes zoster (Infections and infestations) | 2
Infected skin ulcer (Infections and infestations) | 2
Influenza (Infections and infestations) | 2
Infusion site infection (Infections and infestations) | 1
Lower respiratory tract infection (Infections and infestations) | 3
Nasopharyngitis (Infections and infestations) | 3
Oral fungal infection (Infections and infestations) | 1
Oral herpes (Infections and infestations) | 1
Pharyngitis (Infections and infestations) | 1
Respiratory tract infection (Infections and infestations) | 2
Rhinitis (Infections and infestations) | 1
Sinusitis (Infections and infestations) | 1
Tonsillitis (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 4
Viral infection (Infections and infestations) | 1
Vulvovaginal candidiasis (Infections and infestations) | 2
Back injury (Injury, poisoning and procedural complications) | 1
Contusion (Injury, poisoning and procedural complications) | 1
Joint injury (Injury, poisoning and procedural complications) | 1
Procedural site reaction (Injury, poisoning and procedural complications) | 1
Wound necrosis (Injury, poisoning and procedural complications) | 1
Alanine aminotransferase increased (Investigations) | 1
Aspartate aminotransferase increased (Investigations) | 2
Blood albumin decreased (Investigations) | 1
Blood alkaline phosphatase increased (Investigations) | 1
Blood amylase increased (Investigations) | 1
Blood cholesterol increased (Investigations) | 1
Blood creatine phosphokinase increased (Investigations) | 3
Blood triglycerides increased (Investigations) | 2
Blood urea increased (Investigations) | 1
Blood uric acid decreased (Investigations) | 1
C-reactive protein increased (Investigations) | 3
Electrocardiogram QRS complex abnormal (Investigations) | 1
Electrocardiogram abnormal (Investigations) | 1
Gamma-glutamyltransferase increased (Investigations) | 3
Haematocrit decreased (Investigations) | 1
Haemoglobin decreased (Investigations) | 1
Heart rate irregular (Investigations) | 1
High density lipoprotein decreased (Investigations) | 1
Laboratory test interference (Investigations) | 1
Lipase increased (Investigations) | 1
Neutrophil count decreased (Investigations) | 1
Platelet count increased (Investigations) | 1
Protein total abnormal (Investigations) | 1
Red blood cell count decreased (Investigations) | 1
Red blood cell sedimentation rate increased (Investigations) | 4
Troponin I increased (Investigations) | 2
Weight decreased (Investigations) | 2
Weight increased (Investigations) | 1
White blood cell count decreased (Investigations) | 3
Decreased appetite (Metabolism and nutrition disorders) | 3
Dehydration (Metabolism and nutrition disorders) | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1
Iron deficiency (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 7
Back pain (Musculoskeletal and connective tissue disorders) | 1
Groin pain (Musculoskeletal and connective tissue disorders) | 1
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 1
Joint stiffness (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3
Sensation of heaviness (Musculoskeletal and connective tissue disorders) | 1
Systemic sclerosis (Musculoskeletal and connective tissue disorders) | 1
Tenosynovitis stenosans (Musculoskeletal and connective tissue disorders) | 1
Dizziness (Nervous system disorders) | 1
Dysgeusia (Nervous system disorders) | 1
Headache (Nervous system disorders) | 5
Hypoaesthesia (Nervous system disorders) | 1
Neuralgia (Nervous system disorders) | 1
Paraesthesia (Nervous system disorders) | 1
Depression (Psychiatric disorders) | 2
Insomnia (Psychiatric disorders) | 2
Sleep disorder (Psychiatric disorders) | 1
Menorrhagia (Reproductive system and breast disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 1
Dry skin (Skin and subcutaneous tissue disorders) | 1
Hypoaesthesia facial (Skin and subcutaneous tissue disorders) | 1
Lentigo (Skin and subcutaneous tissue disorders) | 1
Panniculitis (Skin and subcutaneous tissue disorders) | 1
Periorbital oedema (Skin and subcutaneous tissue disorders) | 5
Pruritus (Skin and subcutaneous tissue disorders) | 9
Rash (Skin and subcutaneous tissue disorders) | 1
Rash generalised (Skin and subcutaneous tissue disorders) | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1
Skin tightness (Skin and subcutaneous tissue disorders) | 3
Skin ulcer (Skin and subcutaneous tissue disorders) | 5
Swelling face (Skin and subcutaneous tissue disorders) | 1
Erythromelalgia (Vascular disorders) | 1
Raynaud's phenomenon (Vascular disorders) | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.